CLINICAL TRIAL: NCT06171009
Title: Brief Mindfulness Intervention for Orthopedic Patients in the Clinic Waiting Room: Mechanistic Investigation
Brief Title: Brief Mindfulness Intervention for Orthopedic Patients: Mechanistic Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00004419
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Coping Information (Active Comparator)
  Interventions: Behavioral: Pain Coping Information
- Mindful Pain Management (Experimental)
  Interventions: Behavioral: Mindful Pain Management

INTERVENTIONS:
Behavioral: Pain Coping Information — A 4-minute audio recording providing common pain coping techniques (e.g., ice, rest, medication, surgery).
  Arms: Pain Coping Information
Behavioral: Mindful Pain Management — A 4-minute audio recording consisting of a 1-minute introduction to mindfulness followed by a 1-minute and 30-second mindful breathing practice and a 1-minute and 30-second mindfulness of pain practice.
  Arms: Mindful Pain Management

SUMMARY:
This is a single-site, two-arm, parallel-group randomized clinical trial (RCT). The analgesic effects of a 4-minute audio-recorded mindfulness intervention for orthopedic patients will be investigated relative to a 4-minute audio-recoding about pain psychoeducation. Analgesic mechanisms of mindfulness will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Seeking treatment at the Tallahassee Orthopedic Center

Exclusion Criteria:

* Cognitive impairment preventing completion of study procedures.
* Other unstable illness judged by medical staff to interfere with study involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Change in Pain Unpleasantness Numeric Rating Scale | Immediately before to after 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most unpleasant pain imaginable.

SECONDARY OUTCOMES:
Change in Pain Intensity Numeric Rating Scale | Immediately before to after 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most intense pain imaginable.
Change in Decentering | Immediately before to after 4-minute audio recording
  Decentering will be measured by the single, decentering item from the state version of the validated Metacognitive Processes of Decentering Scale. This item will be scored with a Likert scale item ranging from 0-10, with higher scores representing greater decentering.
Change in Self-Transcendent State | Immediately before to after 4-minute audio recording
  Self-transcendent state will be measured by the three-item, state version of the validated Nondual Awareness Dimensional Assessment. These three items will be scored with a Likert scale item ranging from 0-10, with higher scores representing greater self-transcendence.

CONTACTS AND LOCATIONS:
Locations (1):
- Tallahassee Orthopedic Clinic (TOC), Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hanley AW, Gibson R, Davis A, Stecher C, Childs K, Worts P. Mindfulness in the Orthopedic Clinic Waiting Room Decreases Pain: Results From A Randomized Controlled Trial. Int J Behav Med. 2025 Nov 10. doi: 10.1007/s12529-025-10398-3. Online ahead of print. PMID 41214294